CLINICAL TRIAL: NCT01123408
Title: Clozapine and Olanzapine in the Treatment of Violence in Schizophrenic Patients
Brief Title: Clozapine and Olanzapine Treatment of Aggression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Responsible Party: Krakowski, Menahem, Nathan Kline Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2244
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Schizophrenia
Keywords: schizophrenia; aggression; clozapine; olanzapine
MeSH Terms: conditions — Schizophrenia; Aggression | interventions — Clozapine; Olanzapine; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- clozapine (Experimental): During the first 6 weeks clozapine was gradually increased to 500 mg/day and then continued. For the next period, it could vary from 200-800 mg/day;
  Interventions: Drug: Clozapine
- Olanzapine (Experimental): During the first 6 weeks olanzapine was increased to 20 mg and remained fixed for until the end of six week. During the last 6 weeks olanzapine could vary from 10 to 30 mg/day
  Interventions: Drug: Olanzapine
- Haloperidol (Active Comparator): During the first 6 weeks haloperidol was increased to 20 mg and remained fixed for until the end of six week. During the last 6 weeks the dose could vary from 10 to 30 mg/day
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Clozapine — 500 mg/day
  Other Names: clozaryl
  Arms: clozapine
Drug: Olanzapine — 20 mg/day
  Other Names: zyprexa
  Arms: Olanzapine
Drug: Haloperidol — 20 mg/day
  Other Names: Haldol
  Arms: Haloperidol

SUMMARY:
This was a double-blind randomized study with three treatment arms: clozapine, olanzapine and haloperidol. We compared these three medications in the treatment of aggressive behavior over a 12 week period.

DETAILED DESCRIPTION:
Objective: The purpose of our study was the investigation of the effect of atypical antipsychotic agents on interpersonal violence and aggression.

We compared the efficacy of two atypical antipsychotic agents, clozapine and olanzapine with one another and with haloperidol in the treatment of physical assaults and other assaultive behaviors in physically assaultive patients with schizophrenia and schizoaffective disorder.

Method: The subjects were 110 physically assaultive inpatients diagnosed with schizophrenia or schizoaffective disorder.

They were randomly assigned to treatment with clozapine (N=37), olanzapine (N=37) or haloperidol (N=36) in a 12-week, double-blind trial. Incidents of overt aggression were recorded and their severity was scored with the Modified Overt Aggression Scale (MOAS). Psychiatric symptoms were assessed through the Positive and Negative Syndrome Scale (PANSS). We also assessed various side effects and monitored vital signs and drew bloods.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 60 years.
* Diagnosis of schizophrenia or schizoaffective disorder.
* Aggression: One episode of physical assault directed at another person in the hospital and persistence of violence/hostility for two weeks, as evidenced by the presence of some other physical, verbal or property assault or hostility, which would result in a score of 4 or more on the Positive and Negative Syndrome Scale (PANSS) Hostility Item.

Exclusion Criteria:

* Patients who were hospitalized for more than a year
* Patients who had a history of nonresponse to clozapine, olanzapine or haloperidol (defined as a lack of improvement despite a contiguous adequate trial of medication)
* Patients who had a history of clozapine, olanzapine, or haloperidol intolerance
* Patients who had medical conditions that would be adversely affected by any of these three medications.
* Patients who received a depot antipsychotic within 30 days before randomization.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 1999-06; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Number of aggressive incidents | 12 weeks
  The Modified Overt Aggression scale (MOAS) was used to record all aggressive incidents. The primary measure was the total score on the MOAS as well as the score on the MOAS physical aggression subscale

SECONDARY OUTCOMES:
Psychiatric Symptoms | 12 weeks
  Psychiatric symptoms were assessed with the Positive and Negative Syndrome Scale (PANSS) weekly for the first 4 weeks and then bi-weekly for the remainder of the study
Side effects of medications | 12 weeks
  The side effects of the medications were measured with the ESRS on a weekly basis for the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bennett L Leventhal, MD, Study Director — Nathan Kline Institute
Locations (1):
- Nathan Kline Institute, Orangeburg, New York, United States

REFERENCES:
- [Result] Krakowski MI, Czobor P, Citrome L, Bark N, Cooper TB. Atypical antipsychotic agents in the treatment of violent patients with schizophrenia and schizoaffective disorder. Arch Gen Psychiatry. 2006 Jun;63(6):622-9. doi: 10.1001/archpsyc.63.6.622. PMID 16754835
- [Result] Krakowski MI, Czobor P, Nolan KA. Atypical antipsychotics, neurocognitive deficits, and aggression in schizophrenic patients. J Clin Psychopharmacol. 2008 Oct;28(5):485-93. doi: 10.1097/JCP.0b013e3181855cd6. PMID 18794642
- [Derived] Ibragimov K, Keane GP, Carreno Glaria C, Cheng J, Llosa AE. Haloperidol (oral) versus olanzapine (oral) for people with schizophrenia and schizophrenia-spectrum disorders. Cochrane Database Syst Rev. 2024 Jul 3;7(7):CD013425. doi: 10.1002/14651858.CD013425.pub2. PMID 38958149
- [Derived] Krakowski M, Tural U, Czobor P. The Importance of Conduct Disorder in the Treatment of Violence in Schizophrenia: Efficacy of Clozapine Compared With Olanzapine and Haloperidol. Am J Psychiatry. 2021 Mar 1;178(3):266-274. doi: 10.1176/appi.ajp.2020.20010052. Epub 2021 Jan 21. PMID 33472389
- [Derived] Krakowski MI, Czobor P. Executive function predicts response to antiaggression treatment in schizophrenia: a randomized controlled trial. J Clin Psychiatry. 2012 Jan;73(1):74-80. doi: 10.4088/JCP.11m07238. Epub 2011 Nov 29. PMID 22152404